CLINICAL TRIAL: NCT03730714
Title: Surgicel; a Probable Analgesic Reservoir for Post-laparoscopic Cholecystectomy Pain Management; Randomized Controlled Double-blind Trial
Brief Title: Surgicel and Analgesic Reservoir
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esam Hamed, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Surgicel
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local; Epinephrine; Morphine; Surgicel; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ggroup LAM (Active Comparator): Patients will receive local anesthesia Bupivacaine 0.5% 20 ml (no more than 2 mg/kg) plus lidocaine 2% 10 ml (no more than 3 mg/kg) mixed together, plus epinephrine 5 mcg/ml (max 150 mcg), combined with morphine 0.1 mg/kg (max10 mg) instilled into the assigned areas according to the technique.
  Interventions: Drug: "Local Anesthetic", "Epinephrine" and "Morphine"
- Ggroup LAMG (Active Comparator): Patients will receive the same mixture in LAM-group to soak the surgicel according to the previous planned technique.
  Interventions: Drug: "Local Anesthetic", "Epinephrine", "Morphine" and "Surgicel"
- Group CG (Active Comparator): Patients will receive normal saline 0.9% to soak the surgicel according to the planned technique.
  Interventions: Drug: "Normal Saline"

INTERVENTIONS:
Drug: "Local Anesthetic", "Epinephrine" and "Morphine" — local anesthesia Bupivacaine 0.5% 20 ml (no more than 2 mg/kg) plus lidocaine 2% 10 ml (no more than 3 mg/kg) mixed together, plus epinephrine 5 mcg/ml (max 150 mcg), combined with morphine 0.1 mg/kg (max10 mg)
  Arms: Ggroup LAM
Drug: "Local Anesthetic", "Epinephrine", "Morphine" and "Surgicel" — Surgicel soaked with mixture of: local anesthesia Bupivacaine 0.5% 20 ml (no more than 2 mg/kg) plus lidocaine 2% 10 ml (no more than 3 mg/kg) mixed together, plus epinephrine 5 mcg/ml (max 150 mcg), combined with morphine 0.1 mg/kg (max10 mg)
  Arms: Ggroup LAMG
Drug: "Normal Saline" — normal saline 0.9% to soak the surgicel according to the planned technique
  Arms: Group CG

SUMMARY:
Laparoscopic cholecystectomy (LC) is a widespread surgical procedure with superior outcomes in terms of the incurred postoperative pain, recovery time, cosmetic, and morbidity issues. Although it is associated with less postoperative pain compared to open cholecystectomy, but patients still experience significant pain. Pain after LC is categorized into three types: referred pain to the right shoulder due to diaphragmatic stretching during gas insufflation; visceral pain due to dissection and injury at the hepatic fossa during gall bladder removal; and somatic pain due to tissue injury at the port sites. Since the discovery of LC in 1987 by a French surgeon, Phillipe Mouret, it became the gold standard for surgical excision of the gallbladder. Local anesthetics (LA) has been tried for analgesia after LC in variable techniques and concentrations. It was proved to be a safe and valid method for reducing pain after LC instilled intraperitoneal and infiltrated at the port sites.

Surgicel is an absorbable gelatin sponge that is non-toxic, non-allergenic, non-immunogenic, and non-pyrogenic. It is gamma-sterilized and provided with double packing. The sponge is easily cut to fit the surgical cavity. It may be applied dry to the wound. It absorbs 40 times its weight of whole blood or 50 times of water and adheres easily to the bleeding site. It forms a stable adherent coagulum. When implanted in vivo, it is completely absorbed within 3-5 weeks. The rationale for using this sponge as interposition material is to act as a carrier for the analgesic drugs and allow for its local sustained release, and for local hemostasis. Bupivacaine will be used as the main local anesthetic medication in the study. It provides variable pain relief when either used to irrigate intraperitoneal space as a sole analgesic or combined with opioids. Lidocaine 2% will be mixed with bupivacaine to expedite the onset of analgesia. Epinephrine will be used as 5 microgram/ml of the total mixture of used fluids in order to prolong the time of action of the block.

DETAILED DESCRIPTION:
Eligibility and type of the study: This prospective randomized placebo-controlled double-blind study will be conducted after approval from the Institutional Ethics Committee and obtaining a written informed consent from patients undergoing elective laparoscopic cholecystectomy under general anesthesia.

Sample Size: Sample size was calculated according to the previously conducted similar studies in the same field. Based on a pilot study, where the incidence of postoperative pain after laparoscopies was found to be more than 70% and intervention that can cause 50% reduction in this incidence was required. With a power of 90% and type I error of 5%, 26 patients were required to be in each group but to avoid possible patients dropouts, the number of patients in each group is increased to 30 (total of 90 patients).

Drugs Coding and Randomization: Patients will be randomly allocated into three equal groups (30 patients each) using a computer-generated table of random numbers in order to allocate the patients into the three study groups. Neither the anesthesia provider nor the participant will be aware of the study group or the drug used. One anesthesiologist (not included in the procedure, observation or in the data collection) will prepare the study drugs. Two surgeons with average similar level of experience in the field will operate upon patients sequentially without a specific order. All patients will have full explanation about the anesthetic and analgesic techniques they will have before signing their consent.

Anesthesia Technique:

* Before the day of the surgery, patients will visit the outpatient clinic for medical assessment and description of the study protocol after securing their eligibility to participate in the study. Laboratory investigations will be performed and patients will sign the consent. All patients will receive the standard general anesthesia technique followed in the hospital: preoperative 8 hours of NPO, premedication with proton pump inhibitor and antiemetic.
* At operative theatre, patients will be connected to five standard monitoring measures: electrocardiography (ECG), non-invasive blood pressure (NIBP), pulse oxymetry (SpO2), core body temperature, and end-tidal carbon dioxide. An intravenous cannula 18G will be inserted in the dorsum of the non-dominant hand and normal saline 0.9% IV fluids will be infused at a rate of (6-8 ml/kg/h) throughout the surgery.
* After 3 minutes of pre-oxygenation with 100% O2 via the appropriate size face mask, general anesthesia will be induced with 1 µg/kg of fentanyl, 2-3 mg/kg of propofol, cisatracurium (0.15 mg/kg). Patients will be intubated with an appropriate size cuffed endotracheal tube under direct laryngoscopy after complete muscular relaxation. Anesthesia will be maintained with sevoflurane at 2-3% MAC and cisatracurium 0.03 mg/kg. Mechanical ventilation will be maintained and respiratory parameters will be adjusted to keep the end-tidal CO2 at 35-45 mmHg. At the end of the surgery, residual neuromuscular blockade will be pharmacologically reversed using neostigmine 0.04 mg/kg and atropine 0.02 mg/kg, and trachea will be extubated once the patient is showing clinical signs of clearance from neuromuscular blockade and TOF ratio of 0.9 is achieved. In order to control postoperative pain; the patients will receive I.V. paracetamol 1 gm (Perfalgan, Paracetamol 1000 mg. UPSA laboratories, France).

The Study Technique:

After the end of the operative procedure, the patient will have a cut piece of surgicel folded, passed through the big port and intersected dry to cover the gallbladder bed area of the hepatic fossa. The prepared study mixture of medicine will be 32 ml:

* Instilled to soak the surgicel at the hepatic fossa (10 ml).
* Splash the undersurface of the right copula of the diaphragm (10 ml).
* Instilled to soak small pieces of surgicel intersected in the port areas (12 ml).

Groups:

1. First study group (LAM) will receive local anesthesia Bupivacaine 0.5% 20 ml (no more than 2 mg/kg) plus lidocaine 2% 10 ml (no more than 3 mg/kg) mixed together, plus epinephrine 5 mcg/ml (max 150 mcg), combined with morphine 0.1 mg/kg (max10 mg) instilled into the assigned areas according to the technique.
2. Second study group (LAMG) will receive the same mixture in LAM-group to soak the surgicel according to the previous planned technique
3. Control group (CG) will receive normal saline 0.9% to soak the surgicel according to the planned technique

Statistical Analysis:

Data will be collected and analyzed by computer program SPSS (SPSS Inc., Chicago, Illinos, USA) version 23. Data will be expressed as means, standard deviations, ranges, numbers and percentages. The analysis of variance and Chi-square test will be used to assess that the study groups are matched in terms of demographic data. Chi-Square or Fisher exact test will be used to determine significance for categorical variables. T-test or Mann-Whitney test if necessary will be used to determine significance for numeric variables. Kruskal-Wallis test followed by the Wilcoxon matched pairs rank test; will be used specifically to compare VAS and VRS. P value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old patients from both genders scheduled for laparoscopic cholecystectomy
* Clinical and laboratory multisystem preoperative evaluation prove a health status of American society of Anesthesiology grade I/II
* Absence of current active inflammatory medical condition

Exclusion Criteria:

* Allergic reaction to the study medicine
* Patients' health status beyond the specified range
* Patients with seizure diseases
* Patients with significant chronic respiratory disease
* Patients with intraperitoneal infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Visual Analouge Scale | 24 hours
  Postoperative abdominal and shoulder pain using 0-10 scale (with 0 indicating no pain and 10 as the most severe pain ever experienced)

SECONDARY OUTCOMES:
Peak expiratory flow rate | 60 minutes
  by peak flow meter; a portable, inexpensive, hand-held device used to measure how air flows from the lungs in one fast blast.
Postoperative Complications | 24 hours
  Percentages of patients with any postoperative complications will be recorded and treated promptly.
5-point Likert scale | 24 hours
  Patient satisfaction score: (1= very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Esam A. Hamed, M.D., Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided